CLINICAL TRIAL: NCT02027831
Title: Near-infrared Fluorescence Imaging During Neck Dissection in Head and Neck Cancer Patients After Intravenous Injection of Indocyanine Green (a Feasibility Study)
Brief Title: NIR Fluorescence Imaging During Neck Dissection in Head and Neck Cancer Patients After iv Injection of ICG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HN-ICG-IV
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Head and Neck Cancer
Keywords: lymph nodes
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indocyanine Green (Experimental): Intravenous injection of 0,25 mg/kg Indocyanine Green
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green
  Other Names: ICG

SUMMARY:
The purpose of this study is to determine if NIR fluorescent imaging is an effective approach to detect the margins of head and neck tumours or lymph nodes draining the tumour

DETAILED DESCRIPTION:
Primary objective:

definition of the distribution of intravenously injected ICG in the normal and pathological lymph nodes draining the dissected tumor in head and neck cancer patients or in nodes recurrences in head and neck cancer

Secondary objectives:

* Evaluation of the ability of NIR fluorescence imaging to determine the tumoral volume, specifically the margins of the tumoral tissues (in the operating room and in the pathology department)
* Analysis of the correlation between ICG fluorescence and tumoral invasion in the dissected lymph nodes

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring neck dissection with or without resection of the primary (the decision and the type of neck dissection are preliminary decided during head and neck multidisciplinary oncologic consultation).
* Informed consent form signed.

Exclusion Criteria:

* Age less than18 years old.
* Inability to give informed consent.
* History of allergy or hypersensitivity against the investigational product (its active substance or ingredients), to iodine or to shellfish.
* Apparent hyperthyroidism, autonomous thyroid adenoma, unifocal, multifocal or disseminated autonomies of the thyroid gland.
* Documented coronary disease.
* Advanced renal impairment (creatinine > 1,5mg/dl).
* During the 2 weeks before the enrolment, concurrent medication which reduces or increases the extinction of ICG (i.e. anticonvulsants, haloperidol and Heparin).
* Pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the capacity of ICG to detect cervical lymph nodes after IV injection | 7 months
  After IV injection of Indocyanine Green just before the surgery to head and neck cancer patients, we will study the fluorescence due to ICG in cervical lymph nodes and in the primary lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Digonnet, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Brussels Capital, Belgium